CLINICAL TRIAL: NCT00541047
Title: Radiation Therapy and Androgen Deprivation Therapy in Treating Patients Who Have Undergone Surgery for Prostate Cancer (RADICALS)
Brief Title: RADICALS - Radiotherapy and Androgen Deprivation In Combination After Local Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Principal Investigator, Cheryl Pugh, Clinical Project Manager, University College, London
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000571528; MRC-RADICALS-PR10 (Other: MRC at UCL); ISRCTN40814031 (Registry Identifier: ISRCTN); 2006-000205-34 (EudraCT Number); NCT00541047 (Other: NCT); 00316/0223/001-0001 (Other: CTA); PR13 (Other Grant/Funding Number: Canadian Cancer Society - Research Institute)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Complications; Prostate Cancer; Sexual Dysfunction; Urinary Complications
Keywords: sexual dysfunction; urinary complications; gastrointestinal complications; adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological | interventions — bicalutamide; Goserelin; Leuprolide; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- RADICALS-RT: Early RT (Experimental)
  Interventions: Procedure: adjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy
- RADICALS-RT: Salvage RT (Experimental)
  Interventions: Procedure: adjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy
- RADICALS-HD: Radiotherapy Alone (Experimental)
  Interventions: Procedure: adjuvant therapy; Radiation: radiation therapy
- RADICALS-HD: Radiotherapy + 6 months (Experimental)
  Interventions: Drug: bicalutamide; Drug: goserelin acetate; Drug: leuprolide acetate; Procedure: adjuvant therapy; Radiation: radiation therapy
- RADICALS-HD: Radiotherapy + 24 months (Experimental)
  Interventions: Drug: bicalutamide; Drug: goserelin acetate; Drug: leuprolide acetate; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide
  Arms: RADICALS-HD: Radiotherapy + 24 months; RADICALS-HD: Radiotherapy + 6 months
Drug: goserelin acetate
  Arms: RADICALS-HD: Radiotherapy + 24 months; RADICALS-HD: Radiotherapy + 6 months
Drug: leuprolide acetate
  Arms: RADICALS-HD: Radiotherapy + 24 months; RADICALS-HD: Radiotherapy + 6 months
Procedure: adjuvant therapy
Procedure: quality-of-life assessment
  Arms: RADICALS-RT: Early RT; RADICALS-RT: Salvage RT
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Androgens can cause the growth of prostate cancer cells. Androgen deprivation therapy, such as goserelin, leuprolide, or bicalutamide, may lessen the amount of androgens made by the body. Giving radiation therapy together with androgen deprivation therapy may kill more prostate cancer cells.

PURPOSE: This randomized phase III trial is studying how well giving radiation therapy together with androgen deprivation therapy works in treating patients who have undergone surgery for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the timing of radiotherapy and the use of hormone therapy in conjunction with post-operative radiotherapy.
* Determine the impact of radiotherapy on general quality of life, sexual function, urinary function, and bowel function.
* Determine the impact of duration of hormone therapy on general quality of life and sexual function.

OUTLINE: This is a multicenter study. Patients requiring immediate radiotherapy (RT) are assigned to arm I; patients do not require immediate RT are assigned to arm II. Patients for whom the need of immediate post-operative radiotherapy are uncertain undergo radiotherapy timing randomization within 3 months after surgery and are randomized to 1 of 2 radiotherapy arms.

* Arm I (immediate RT): Within 2 months after randomization, patients undergo radiotherapy to the prostate bed once a day, 5 days a week, for 4 (20 fractions total) or 6.5 weeks (33 fractions total). They may also undergo radiotherapy to the pelvic lymph nodes once a day, 5 days a week, for 4.5 weeks (23 fractions total) at the investigator's discretion.
* Arm II (early salvage RT in case of PSA failure): Within 2 months of confirmation of post-operative biochemical failure, patients undergo radiotherapy as in arm I.

Patients undergoing immediate RT and patients who eventually need early salvage RT undergo hormone therapy duration randomization before the administration of post-operative radiotherapy. Patients are randomized to 1 of 3 hormone therapy arms.

* Arm III (no hormone therapy): Patients do not receive hormone therapy. They receive post-operative RT alone as described above in arm I or II.
* Arm IV (RT and short-term hormone therapy): Beginning approximately 2 months prior to the start of RT, patients receive hormone therapy for 6 months. Hormone therapy* may comprise of LHRH agonist (gonadotrophin-releasing hormone analogue [GnRHa] [e.g., goserelin or leuprolide acetate]) or bicalutamide daily.
* Arm V (RT and long-term hormone therapy): Beginning approximately 2 months prior to the start of RT, patients receive hormone therapy for 24 months. Hormone therapy* may comprise of LHRH agonist (gonadotrophin-releasing hormone analogue [GnRHa] [e.g., goserelin or leuprolide acetate]) or bicalutamide daily.

NOTE: *For Canadian patients, hormonal therapy will consist of LHRH analog (leuprolide acetate) therapy only.

Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed using self-administered questionnaires at baseline and 1, 5, and 10 years after randomization. Health economics information is also collected via patient-administered questionnaires (EQ-5D) at baseline and at 1, 5 and 10 years after randomization.

After completion of study treatment, patients are followed for 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of nonmetastatic adenocarcinoma of the prostate
* Must have undergone radical prostatectomy
* Post-operative serum prostate-specific antigen (PSA) < 0.4 ng/mL
* No post-operative biochemical failure, defined as EITHER two consecutive rises in PSA and final PSA > 0.1 ng/mL OR three consecutive rises in PSA (for patients undergoing hormone therapy duration randomization)

Exclusion criteria:

* Known distant metastases from prostate cancer
* PSA > 5 ng/mL at the time of hormone randomization (for patients undergoing hormone therapy duration randomization)

PATIENT CHARACTERISTICS:

* No other active malignancy likely to interfere with protocol treatment or follow-up

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* Co-enrollment to other trials is permitted, providing this does not interfere with the outcome measures
* 5-α reductase inhibitors, soya, selenium, and vitamin E are acceptable non-trial therapies

Exclusion criteria:

* Prior hormone therapy
* Bilateral orchidectomy
* Prior pelvic radiotherapy
* Neoadjuvant treatment
* Other concurrent therapies for prostate cancer (e.g., estrogens or cytotoxic chemotherapy) prior to disease progression

Ages: 0 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4236 (Actual)
Dates: Start 2007-11; Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Disease-specific survival (i.e., death due to prostate cancer) (RADICALS-HD) | up 12 years
Freedom from distant metastases (any distance metastases or prostate cancer death) (RADICALS-RT) | up 12 years

SECONDARY OUTCOMES:
Freedom from treatment failure | up 12 years
Clinical progression-free survival | up 12 years
Overall survival | up 12 years
Non-protocol hormone therapy | up 12 years
Treatment toxicity | up 12 years
Patient reported outcomes - EQ5D | up 12 years
Freedom from biochemical progression (RADICALS-RT) | up 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Parker, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (58):
- Canada (5):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- United Kingdom (53):
  - William Harvey Hospital, Ashford, England
  - North Devon District Hospital, Barnstaple, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Southmead Hospital, Bristol, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Walsgrave Hospital, Coventry, England
  - Mid Cheshire Hospitals Trust- Leighton Hopsital, Crewe, England
  - Mayday University Hospital, Croydon, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Dorset County Hospital, Dorchester, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Princess Alexandra Hospital, Harlow, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Lincoln County Hospital, Lincoln, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - University College Hospital, London, England
  - Guy's Hospital, London, England
  - Royal Marsden - London, London, England
  - Maidstone Hospital, Maidstone, England
  - Clatterbridge Centre for Oncology, Manchester, England
  - Christie Hospital, Manchester, England
  - James Cook University Hospital, Middlesbrough, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Queen's Hospital, Romford, England
  - Rotherham General Hospital, Rotherham, England
  - Hope Hospital, Salford, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Stepping Hill Hospital, Stockport, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Royal Marsden - Surrey, Sutton, England
  - Torbay Hospital, Torquay, England
  - Hillingdon Hospital, Uxbridge, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Cancer Care Centre at York Hospital, York, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ayr Hospital, Ayr, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Glan Clwyd Hospital, Bodelwyddan, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Royal Gwent Hospital, Newport, Wales

IPD SHARING:
Plan to Share IPD: No
Data can be shared on request via emailing mrcctu.radical@ucl.ac.uk

REFERENCES:
- [Result] Parker CC, Clarke NW, Catton C, Kynaston H, Cook A, Cross W, Davidson C, Goldstein C, Logue J, Maniatis C, Petersen PM, Neville P, Payne H, Persad R, Pugh C, Stirling A, Saad F, Parulekar WR, Parmar MKB, Sydes MR. RADICALS-HD: Reflections before the Results are Known. Clin Oncol (R Coll Radiol). 2022 Sep;34(9):593-597. doi: 10.1016/j.clon.2022.06.004. Epub 2022 Jul 6. No abstract available. PMID 35810050
- [Result] Parker CC, Clarke NW, Cook AD, Kynaston HG, Petersen PM, Catton C, Cross W, Logue J, Parulekar W, Payne H, Persad R, Pickering H, Saad F, Anderson J, Bahl A, Bottomley D, Brasso K, Chahal R, Cooke PW, Eddy B, Gibbs S, Goh C, Gujral S, Heath C, Henderson A, Jaganathan R, Jakobsen H, James ND, Kanaga Sundaram S, Lees K, Lester J, Lindberg H, Money-Kyrle J, Morris S, O'Sullivan J, Ostler P, Owen L, Patel P, Pope A, Popert R, Raman R, Roder MA, Sayers I, Simms M, Wilson J, Zarkar A, Parmar MKB, Sydes MR. Timing of radiotherapy after radical prostatectomy (RADICALS-RT): a randomised, controlled phase 3 trial. Lancet. 2020 Oct 31;396(10260):1413-1421. doi: 10.1016/S0140-6736(20)31553-1. Epub 2020 Sep 28. PMID 33002429
- [Result] Vale CL, Fisher D, Kneebone A, Parker C, Pearse M, Richaud P, Sargos P, Sydes MR, Brawley C, Brihoum M, Brown C, Chabaud S, Cook A, Forcat S, Fraser-Browne C, Latorzeff I, Parmar MKB, Tierney JF; ARTISTIC Meta-analysis Group. Adjuvant or early salvage radiotherapy for the treatment of localised and locally advanced prostate cancer: a prospectively planned systematic review and meta-analysis of aggregate data. Lancet. 2020 Oct 31;396(10260):1422-1431. doi: 10.1016/S0140-6736(20)31952-8. Epub 2020 Sep 28. PMID 33002431
- [Derived] Parker CC, Clarke NW, Cook AD, Kynaston H, Catton CN, Cross WR, Petersen PM, Persad RA, Saad F, Bower LC, Logue J, Payne H, Forcat S, Goldstein C, Murphy C, Anderson J, Barkati M, Bottomley DM, Branagan J, Choudhury A, Chung PWM, Cogley L, Goh CL, Hoskin P, Khoo V, Malone SC, Masters L, Morris SL, Nabid A, Ong AD, Raman R, Tarver KL, Tree AC, Worlding J, Wylie JP, Zarkar AM, Parulekar WR, Parmar MKB, Sydes MR; RADICALS investigators. Adding 6 months of androgen deprivation therapy to postoperative radiotherapy for prostate cancer: a comparison of short-course versus no androgen deprivation therapy in the RADICALS-HD randomised controlled trial. Lancet. 2024 Jun 1;403(10442):2405-2415. doi: 10.1016/S0140-6736(24)00548-8. Epub 2024 May 16. PMID 38763154
- [Derived] Parker CC, Kynaston H, Cook AD, Clarke NW, Catton CN, Cross WR, Petersen PM, Persad RA, Pugh CA, Saad F, Logue J, Payne H, Bower LC, Brawley C, Rauchenberger M, Barkati M, Bottomley DM, Brasso K, Chung HT, Chung PWM, Conroy R, Falconer A, Ford V, Goh CL, Heath CM, James ND, Kim-Sing C, Kodavatiganti R, Malone SC, Morris SL, Nabid A, Ong AD, Raman R, Rodda S, Wells P, Worlding J, Parulekar WR, Parmar MKB, Sydes MR; RADICALS investigators. Duration of androgen deprivation therapy with postoperative radiotherapy for prostate cancer: a comparison of long-course versus short-course androgen deprivation therapy in the RADICALS-HD randomised trial. Lancet. 2024 Jun 1;403(10442):2416-2425. doi: 10.1016/S0140-6736(24)00549-X. Epub 2024 May 16. PMID 38763153
- [Derived] Parker CC, Petersen PM, Cook AD, Clarke NW, Catton C, Cross WR, Kynaston H, Parulekar WR, Persad RA, Saad F, Bower L, Durkan GC, Logue J, Maniatis C, Noor D, Payne H, Anderson J, Bahl AK, Bashir F, Bottomley DM, Brasso K, Capaldi L, Chung C, Cooke PW, Donohue JF, Eddy B, Heath CM, Henderson A, Henry A, Jaganathan R, Jakobsen H, James ND, Joseph J, Lees K, Lester J, Lindberg H, Makar A, Morris SL, Oommen N, Ostler P, Owen L, Patel P, Pope A, Popert R, Raman R, Ramani V, Roder A, Sayers I, Simms M, Srinivasan V, Sundaram S, Tarver KL, Tran A, Wells P, Wilson J, Zarkar AM, Parmar MKB, Sydes MR; RADICALS investigators. Timing of radiotherapy (RT) after radical prostatectomy (RP): long-term outcomes in the RADICALS-RT trial (NCT00541047). Ann Oncol. 2024 Jul;35(7):656-666. doi: 10.1016/j.annonc.2024.03.010. Epub 2024 Apr 5. PMID 38583574